CLINICAL TRIAL: NCT04316325
Title: Medical Abortion Via Telemedicine for Women and Adolescents in Moldova
Status: Completed | Type: Observational
Sponsor: Reproductive Health Training Center of the Republic of Moldova (Other)
Collaborators: Grand Challenges Canada (Other); Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: POC-OPT-1902-31934
Record Dates: First submitted 2020-03-18; First posted 2020-03-20 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women and girls seeking abortion.
  Interventions: Drug: Medical abortion

INTERVENTIONS:
Drug: Medical abortion — Trained abortion providers will counsel participants about medical abortion via videoconference or telephone, the abortion medications will be sent to the participants via mail or will be accessed at a pharmacy, the provider will follow up one week later with the participants to assess outcomes, and four weeks later the participant will take a pregnancy test to confirm completion of the abortion

SUMMARY:
This study evaluates the safety, feasibility, and acceptability of a novel medical abortion via telemedicine service in the Republic of Moldova.

DETAILED DESCRIPTION:
Women and girls in Moldova, especially those in rural areas, must travel to regional medical centers to obtain an abortion from a certified gynecologist. This creates barriers to accessing safe abortion that disproportionately affect poor women and girls, through wage loss due to missed work and accrued costs due to transportation. This innovation is a novel service delivery model that allows self-management of medical abortion (MA) with remote guidance from a provider. After confirming their pregnancy, women seeking MA will receive counseling from a gynecologist via videoconference and will subsequently obtain the necessary medication via mail or at at participating pharmacy with prescription. Follow-up will occur 1 weeks later via phone/videoconference (with referral to a doctor if necessary) to confirm MA success and assess the patient's and provider's satisfaction with the service. We hope to demonstrate the feasibility, effectiveness and acceptability of telemedicine MA services in Moldova so that it can thus be integrated into the national public healthcare system. As a result, this project will serve as a model that could be adapted and implemented in nearby countries within the Eastern Europe and Central Asia region.

ELIGIBILITY:
Inclusion Criteria:

* 16 years or older
* Has an unwanted pregnancy
* Confirmed the pregnancy using a test or via ultrasound
* Gestational age of 9 weeks or less
* Has personally decided to end the pregnancy
* Has a device (phone, tablet, or computer) with internet connection, a webcam, and a microphone.
* Has immediate access to emergency services
* Reports no contraindication to medical abortion

Exclusion Criteria:

* Under 16 years of age
* Does not have an unwanted pregnancy
* Did not confirm pregnancy
* Gestational age greater than 9 weeks
* Does not have a device (phone, tablet, or computer) with internet connection, a webcam, and a microphone
* Does not have immediate access to emergency services
* Has an intrauterine device
* Is allergic to abortion medications (mifepristone or misoprostol)
* Has severe anemia or acute porphyria
* Has a condition that affects the ability of blood to clot normally
* Has hepatic failure or chronic renal disease
* Has an ectopic pregnancy
* Has heart disease or other cardiovascular problem
* Has a condition that requires hormone treatment

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women and girls seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 549 (Actual)
Dates: Start 2020-03-20 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Successful termination of pregnancy without adverse events | through study completion, around 15 months
  Percentage of study participants that successfully terminate their pregnancy via the telemedicine medical abortion model without experiencing any adverse events.

SECONDARY OUTCOMES:
Participant satisfaction with the medical abortion via telemedicine service | through study completion, around 15 months
  Percentage of study participants that report being satisfied or very satisfied with the medical abortion via telemedicine service.
Cost savings experienced by study participants | through study completion, around 15 months
  Percentage cost savings among study participants receiving medical abortion via telemedicine in comparison with the cost of in-person medical abortion.
Provider satisfaction | through study completion, around 15 months
  Percentage of medical abortion providers that report being satisfied or very satisfied with the telemedicine service provision process.

CONTACTS AND LOCATIONS:
Overall Officials: Rodica Comendant, MD,PhD, Principal Investigator — Director
Locations (1):
- Reproductive Health Training Center, Chisinau, Moldova